CLINICAL TRIAL: NCT02879656
Title: Non-operative Treatment Versus Surgery With Volar Locking Plate in Treatment of Distal Radius Fracture in 65-year-old and Older Patients - a Prospective, Randomized Controlled Trial
Brief Title: Non-operative Treatment Versus Volar Locking Plate in Treatment of Distal Radius Fracture in Patients Over 65 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Central Finland Hospital District (Other); Satakunta Central Hospital (Other); Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Antti Launonen, MD, PhD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R16105
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Other): Early ustable fracture:
  Phase 1:
  After closed reduction, if satisfactory reduction is not achieved fulfilling the inclusion criteria, the patient is allocated to Cohort 1. The patient is randomized to either non-operative (=Arm 1) or operative treatment (=Arm 2). Patients allocated to non-operative treatment will undergo a standard treatment protocol. Patients allocated to operative treatment will undergo a surgery with volar locking plate with modified Henry's volar approach.
  Interventions: Procedure: non-operative treatment; Procedure: operative treatment
- Cohort 2 (Other): Early stable fracture:
  Phase 1:
  After closed reduction, if satisfactory position is achieved, the patient is allocated to Cohort 2 and conservative treatment is performed as usually.
  Phase 2:
  Patients allocated to Cohort 2, will visit orthopedic outpatient clinic in 1 week in the hospital where the treatment was initially started. If reduction is maintained the patient will undergo standard follow-up visits. If reduction is lost to fulfill the inclusion criteria for surgery the patient is asked to participate to phase 2 of this study. After the patient´s enrollment has been confirmed and informed consent is signed, the patient is randomized to either non-operative (=Arm 3N) or operative treatment (=Arm 3O). If allocated to non-operative treatment patient will undergo the same protocol as those in the Arm 1. Patients allocated to operative treatment will undergo surgery with volar locking plate with standard volar approach.
  Interventions: Procedure: non-operative treatment; Procedure: operative treatment

INTERVENTIONS:
Procedure: non-operative treatment — conservative treatment with 5 weeks cast immobilization
Procedure: operative treatment — surgery with volar locking plate with modified Henry's volar approach

SUMMARY:
The present collaboration study on the treatment of distal radius fractures is aimed to:

(i) to compare non-operative treatment to volar plating in the treatment of initially malaligned distal radius fractures in patients aged 65 and older in terms of functional outcome measured with PRWE

(ii) to compare non-operative treatment to volar plating in the treatment of distal radius fractures with early instability during follow-up, i.e., loss of reduction at 1 week (range 5 to 10 days) in patients aged 65 and older in terms of functional outcome measured with PRWE

(iii)to compare pain, disability, quality of life, grip strength, and the number of complications after non-operative treatment and the initial and delayed operative treatment of distal radius fracture

(iv) to assess the effect of pain catastrophizing score (PCS) on the functional outcome of non-operatively and operatively treated distal radius fracture

(v) to assess the association between physical activity and the number of wrist movements measured with Axivity accelerometer and functional outcome measured with PROMs of non-operatively and operatively treated distal radius fractures

(vi) to assess the effect of initial as well as the final radiological parameters on the functional outcome

(vii) to assess the correlation of probability of radiological malalignment estimated by clinical prediction rule (EWC) with functional outcome measured with PRWE and PASS

ELIGIBILITY:
Inclusion Criteria:

* low energy intra or extra-articular dorsally displaced distal radius fracture within 3 cm of the radiocarpal joint, diagnosed with lateral and posterior-anterior radiographs in ER
* >10° dorsal tilt and/or over 2 mm step-off and/or over 3 mm shortening in the radiograph

Exclusion Criteria:

* Refuse to participate the study
* Open fracture more than Gustilo 1 gradus
* Age under 65 years
* Chauffeure's or Barton´s fracture
* Smith´s fracture (volar angulation of the fracture)
* Does not understand written and spoken guidance in local languages
* Pathological fracture or previous fracture in the same wrist or forearm

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 291 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Change over time in Patient Rated Wrist Evaluation (PRWE) | 3 months, 1 year, 2 years
  PRWE is the primary outcome measure of wrist pain and disability in the study.
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists three subscales: Pain, Function and Cosmetics.

SECONDARY OUTCOMES:
Disability of the wrist measured with the Disability of the Arm, Shoulder and Hand (QuickDASH) questionnaire | 3 months, 1 year, 2 years
  The QuickDASH is self-reported questionnaire and shortened version of DASH outcome measure to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb in 11 dimensions in 1-5 scale.
Quality of life measured with the 15-D | Baseline, 3 months, 1 year, 2 years
  The 15D is a validated, generic, self-administered instrument for assessing the health related quality of life among adults. It combines the advantages of a preference-based and single index measure on a 0-1 scale.
Pain measured in Visual Analogue Scale (VAS) | 3 months, 1 year, 2 years
  The VAS is derived by health care professional question of pain in scale 0 to 10 in which 0 implies no pain and 10 the worst possible pain.
Grip strength measured with a dynamometer | 3 months, 1 year
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in percentage of the uninjured side.
Pain catastrophizing measured with the pain catastrophizing scale (PCS) | baseline, 3 months, 1 year, 2 years
  The pain catastrophizing scale (PCS) is measured with a self-administered questionnaire. The PCS is designed to measure person's willingness to catastrophize the pain while they are experiencing it. In the questionnaire patients answer questions about how they feel and think when they are in pain and it can be taken while they are not experiencing pain.
Physical activity measured with Axivity accelerometer | 3 months, 1 year
  Physical activity will be measured in a subgroup of patients in two separate follow-up time points.
Self-assessment | Baseline, 1 year, 2 years
  Patient's self-assessment questionnaire will be analyzed to find out which parameters are of most importance for the patient.
EWC | Baseline
  Edinbourgh wrist calculator will be used to estimate the propability of loss of reduction during the follow-up.
Frailty | Baseline
  Clinical Frailty Score

CONTACTS AND LOCATIONS:
Overall Officials: Ville Mattila, Prof, Study Director — Tampere University Hospital; Antti Launonen, MD, Principal Investigator — Tampere University Hospital; Minna Laitinen, adjunct prof, Study Chair — Tampere University Hospital; Teemu Hevonkorpi, MD, Study Chair — Tampere University Hospital; Lauri Raittio, MD, Study Chair — Tampere University Hospital; Toni Luokkala, MD, Study Chair — Central Finland Central Hospital; Aleksi Reito, MD, Study Chair — Central Finland Central Hospital; Juha Kukkonen, MD, Study Chair — Satakunta Central Hospital; Li Felländer-Tsai, MD, Study Chair — Karolinska University Hospital
Locations (5):
- Viborg Regional Hospital, Viborg, Denmark
- Finland (3):
  - Jyväskylä Central Hospital, Jyväskylä
  - Pori Central Hospital, Pori
  - Tampere University Hospital, Tampere
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hevonkorpi TP, Launonen AP, Reito A, Schandorff Skjaerbaek M, Li Y, Luokkala T, Kukkonen J, Paloneva J, Kvistgaard Ostergaard H, Fellander-Tsai L, Laitinen MK, Sumrein BO, Mechlenburg I, Mattila VM; as the NITEP Group (Nordic Innovative Trial to Evaluate osteoPorotic fractures). Nonoperative treatment versus volar locking plating for distal radius fracture in patients aged 65 years or older (DRIFT trial): A randomized controlled trial. PLoS Med. 2025 Sep 5;22(9):e1004728. doi: 10.1371/journal.pmed.1004728. eCollection 2025 Sep. PMID 40911648
- [Derived] Hevonkorpi TP, Launonen AP, Raittio L, Luokkala T, Kukkonen J, Reito A, Sumrein BO, Laitinen MK, Mattila VM; NITEP-group. Nordic Innovative Trial to Evaluate OsteoPorotic Fractures (NITEP-group): non-operative treatment versus surgery with volar locking plate in the treatment of distal radius fracture in patients aged 65 and over - a study protocol for a prospective, randomized controlled trial. BMC Musculoskelet Disord. 2018 Apr 5;19(1):106. doi: 10.1186/s12891-018-2019-5. PMID 29621979